CLINICAL TRIAL: NCT03563222
Title: Prospective, Randomized (1:1), Double-Blind, Parallel-Group, Active-Controlled, Multicenter Study to Compare Safety and Efficacy of Smoflipid to Intralipid 20% in Pediatric Patients of 3 Months to 16 Years of Age Requiring Parenteral Nutrition for at Least 90 Days and up to 1 Year
Brief Title: Safety and Efficacy Study to Compare Smoflipid and Intralipid 20% in Pediatric Patients of 3 Months to 16 Years of Age
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Prematurely stopped in agreement with authorities (FDA)
Sponsor: Fresenius Kabi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SMOF-028-CP4
Record Dates: First submitted 2018-06-05; First posted 2018-06-20 (Actual); Results first posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-11

CONDITIONS: Malnutrition, Child
Keywords: Parenteral nutrition; Pediatrics; Malnutrition; Nutritional needs
MeSH Terms: conditions — Child Nutrition Disorders; Hyperphagia; Malnutrition | interventions — SMOFlipid; soybean oil, phospholipid emulsion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Smoflipid (Experimental): Smoflipid is a sterile, nonpyrogenic, white, homogenous lipid emulsion for intravenous infusion. The lipid content of Smoflipid is 0.20 g/mL, and comprises a mixture of soybean oil, medium chain triglycerides, olive oil, and fish oil. Smoflipid is indicated as a source of calories and essential fatty acids for parenteral nutrition when oral or enteral nutrition is not possible, insufficient, or contraindicated.
  The mean essential fatty acid content of Smoflipid is 35 mg/mL linoleic acid (omega-6) and 4.5 mg/mL α-linolenic acid (omega-3).
  Interventions: Drug: Smoflipid
- Intralipid, 20% (Active Comparator): Intralipid 20% is a sterile, non-pyrogenic fat emulsion intended as a source of calories and essential fatty acids. Intralipid 20% is indicated as a source of calories and essential fatty acids for patients requiring parenteral nutrition for extended periods of time and as a source of essential fatty acids for prevention of essential fatty acid deficiency. The major component fatty acids are linoleic acid, oleic acid, palmitic acid, α-linolenic acid and stearic acid.
  Interventions: Drug: Intralipid, 20%

INTERVENTIONS:
Drug: Smoflipid — The study drugs will be infused via a dedicated line for parenteral nutrition (PN) into a central vein using a central venous catheter or a peripherally inserted central catheter.
  The initial rate of infusion should be no more than 0.05 mL/minute for the first 10 to 15 minutes. If no untoward reactions occur, the rate can be changed to permit infusion of 0.5 mL/kg/hour.
  The individual dosage of study drug should be infused at a constant rate for 10 to 24 h/d. The administration flow rate is determined by dividing the volume of study drug by the duration of the infusion. Maximum infusion rate for lipid should not exceed 0.125 g/kg/h lipid.
  Study drug infusions should be given 5 to 7 days per week. Study treatment will last for a minimum of 90 consecutive days and as long as PN is indicated, up to 365 consecutive days. If the indication for PN continues after Study Day 365, PN will continue per normal institution policy.
  Other Names: Smoflipid® Lipid Injectible Emulsion, USP 20%
  Arms: Smoflipid
Drug: Intralipid, 20% — The study drugs will be infused via a dedicated line for parenteral nutrition (PN) into a central vein using a central venous catheter or a peripherally inserted central catheter.
  The initial rate of infusion should be no more than 0.05 mL/minute for the first 10 to 15 minutes. If no untoward reactions occur, the rate can be changed to permit infusion of 0.5 mL/kg/hour.
  The individual dosage of study drug should be infused at a constant rate for 10 to 24 h/d. The administration flow rate is determined by dividing the volume of study drug by the duration of the infusion. Maximum infusion rate for lipid should not exceed 0.125 g/kg/h lipid.
  Study drug infusions should be given 5 to 7 days per week. Study treatment will last for a minimum of 90 consecutive days and as long as PN is indicated, up to 365 consecutive days. If the indication for PN continues after Study Day 365, PN will continue per normal institution policy.
  Other Names: Intralipid® 20% (20% i.v. fat emulsion)
  Arms: Intralipid, 20%

SUMMARY:
Evaluate the safety and efficacy of Smoflipid compared to standard of care lipid emulsion Intralipid 20% administered via a central vein in pediatric patients 3 months to 16 years of age who require parenteral nutrition for at least 90 days and up to 1 year.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 3 months to 16 years of age.
2. Patients who require PN for at least 5 days/week.
3. Patients who receive 60% or more of their total energy requirements as PN at enrollment and who are expected to receive 60% or more of their total energy requirements as PN for at least 90 days.
4. Written informed consent from parent(s) or legal representative(s). If possible, patient assent must also be obtained (according to local law).

Exclusion Criteria:

1. Known hypersensitivity to fish, egg, soybean, or peanut proteins, or to any of the active ingredients or excipients of Smoflipid or Intralipid 20%.
2. Hyperlipidemia or disorders of lipid metabolism characterized by hypertriglyceridemia (serum triglyceride concentration > 250 mg/dL).
3. Inborn errors of amino acid metabolism.
4. Cardiopulmonary instability (including pulmonary edema, cardiac insufficiency, myocardial infarction, acidosis and hemodynamic instability requiring significant vasopressor support).
5. Hemophagocytic syndrome.
6. Liver enzymes (either AST, or ALT, or GGT) exceeding 5 x upper limit of normal range
7. Direct bilirubin ≥ 2.0 mg/dl
8. INR > 2.
9. Any known hepatic condition outside of Intestinal Failure-Associated Liver Disease (IFALD) that will increase direct bilirubin ≥ 2.0 mg/dl.
10. Clinically significant abnormal levels of any serum electrolyte (sodium, potassium, magnesium, calcium, chloride, phosphate).
11. Active bloodstream infection demonstrated by positive blood culture at screening.
12. Severe renal failure including patients on renal replacement therapy.
13. Abnormal blood pH, oxygen saturation, or carbon dioxide.
14. Pregnancy or lactation.
15. Participation in another clinical study.
16. Unlikely to survive longer than 90 days.

Ages: 3 Months to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Rudolph, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Smoflipid: Smoflipid is a sterile, nonpyrogenic, white, homogenous lipid emulsion for intravenous infusion. The lipid content of Smoflipid is 0.20 g/mL, and comprises a mixture of soybean oil, medium chain triglycerides, olive oil, and fish oil. Smoflipid is indicated as a source of calories and essential fatty acids for parenteral nutrition when oral or enteral nutrition is not possible, insufficient, or contraindicated.
  The mean essential fatty acid content of Smoflipid is 35 mg/mL linoleic acid (omega-6) and 4.5 mg/mL α-linolenic acid (omega-3).
  Smoflipid: The study drugs will be infused via a dedicated line for parenteral nutrition (PN) into a central vein using a central venous catheter or a peripherally inserted central catheter.
  The initial rate of infusion should be no more than 0.05 mL/minute for the first 10 to 15 minutes. If no untoward reactions occur, the rate can be changed to permit infusion of 0.5 mL/kg/hour.
  The individual dosage of study drug should be infused at a constant rate for 10 to 24 h/d. The administration flow rate is determined by dividing the volume of study drug by the duration of the infusion. Maximum infusion rate for lipid should not exceed 0.125 g/kg/h lipid.
  Study drug infusions should be given 5 to 7 days per week. Study treatment will last for a minimum of 90 consecutive days and as long as PN is indicated, up to 365 consecutive days. If the indication for PN continues after Study Day 365, PN will continue per normal institution policy.
- Intralipid, 20%: Intralipid 20% is a sterile, non-pyrogenic fat emulsion intended as a source of calories and essential fatty acids. Intralipid 20% is indicated as a source of calories and essential fatty acids for patients requiring parenteral nutrition for extended periods of time and as a source of essential fatty acids for prevention of essential fatty acid deficiency. The major component fatty acids are linoleic acid, oleic acid, palmitic acid, α-linolenic acid and stearic acid.
  Intralipid, 20%: The study drugs will be infused via a dedicated line for parenteral nutrition (PN) into a central vein using a central venous catheter or a peripherally inserted central catheter.
  The initial rate of infusion should be no more than 0.05 mL/minute for the first 10 to 15 minutes. If no untoward reactions occur, the rate can be changed to permit infusion of 0.5 mL/kg/hour.
  The individual dosage of study drug should be infused at a constant rate for 10 to 24 h/d. The administration flow rate is determined by dividing the volume of study drug by the duration of the infusion. Maximum infusion rate for lipid should not exceed 0.125 g/kg/h lipid.
  Study drug infusions should be given 5 to 7 days per week. Study treatment will last for a minimum of 90 consecutive days and as long as PN is indicated, up to 365 consecutive days. If the indication for PN continues after Study Day 365, PN will continue per normal institution policy.
Period: Overall Study
Arm/Group | Smoflipid | Intralipid, 20%
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was prematurely terminated
Groups:
- Total: Total of all reporting groups
Arm/Group | Smoflipid | Intralipid, 20% | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 4 [4 to 4] |  | 4 [4 to 4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body mass index [Mean (Full Range); unit: kg/m²] | 16.34 [16.34 to 16.34] |  | 16.34 [16.34 to 16.34]

OUTCOME MEASURES:

1. Primary Outcome: Body Weight
Description: Body weight of patients (patients < 36 months of age)
Time Frame: from day 1 monthly to day 365
Population: Analysis not perfomed due to early study termination. Single subject's data will not be disclosed to maintain confidentiality.
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Body Height
Description: Height oder length of body (patients <36 months of age)
Time Frame: from day 1 monthly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

3. Primary Outcome: Head Circumference
Description: Circumference of head in patients > 36 months old
Time Frame: from day 1 monthly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

4. Primary Outcome: Fatty Acid Profile in Total Plasma
Description: Fatty acid profile including linoleic acid, α-linolenic acid, arachidonic acid, docosahexaenoic acid, eicosapentaenoic acid and Mead acid, analyzed in total plasma
Time Frame: from day 1 monthly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

5. Primary Outcome: Fatty Acid Profile in Red Blood Cell Membranes
Description: Fatty acid profile including linoleic acid, α-linolenic acid, arachidonic acid, docosahexaenoic acid, eicosapentaenoic acid and Mead acid, analyzed in red blood cell membranes
Time Frame: from day 1 monthly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

6. Primary Outcome: Triene/Tetraene Ratio
Description: Triene/tetraene ratio (Holman Index) in total plasma to assess essential fatty acid deficiency (EFAD)
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

7. Primary Outcome: Number of Patients in Each Treatment Group With Direct Bilirubin Levels > 2 mg/dL
Time Frame: from day 1 monthly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

8. Primary Outcome: Time Until Reaching Direct Bilirubin Levels > 2 mg/dL
Time Frame: from day 1 monthly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

9. Primary Outcome: Sterols in Plasma Including Phytosterols
Time Frame: from day 1 monthly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

10. Primary Outcome: Change From Baseline Triglycerides
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

11. Primary Outcome: Change From Baseline Urea Nitrogen
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

12. Primary Outcome: Change From Baseline Alanine Aminotransferase (ALT)
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

13. Primary Outcome: Change From Baseline Aspartate Aminotransferase (AST)
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

14. Primary Outcome: Change From Baseline Direct Bilirubin
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

15. Primary Outcome: Change From Baseline Total Bilirubin
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

16. Primary Outcome: Change From Baseline Gamma-glutamyl Transferase (GGT)
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

17. Primary Outcome: Change Form Baseline Alkaline Phosphatase (ALP)
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

18. Primary Outcome: Change From Baseline Creatinine
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

19. Primary Outcome: Change From Baseline Electrolytes (Na, K, Mg, Cl,Ca, Phosphate)
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

20. Primary Outcome: Change From Baseline Trace Elements (Ferritin, Zn, Se, Cu, Mn, Cr)
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

21. Primary Outcome: Change From Baseline Glucose
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

22. Primary Outcome: Change From Baseline Total Protein
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

23. Primary Outcome: Change From Baseline C-reactive Protein (CRP)
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

24. Primary Outcome: Change From Baseline White Blood Cell (WBC) Count
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

25. Primary Outcome: Change From Baseline Red Blood Cell (RBC) Count
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

26. Primary Outcome: Change From Baseline Platelet Count
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

27. Primary Outcome: Change From Baseline Hemoglobin
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

28. Primary Outcome: Change From Baseline Hematocrit
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

29. Primary Outcome: Change From Baseline International Normalized Ratio (INR)
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

30. Primary Outcome: Change From Baseline Sterols (Beta-sitosterol, Campesterol, Stigmasterol, Brassicasterol, Ergosterol, Cholesterol, Desmosterol, Lanosterol, Beta-sitostanol, Lathosterol, Squalene)
Time Frame: from day 1 monthly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

31. Primary Outcome: Vital Signs: Blood Pressure
Description: Systolic and diastolic blood pressure
Time Frame: from day 1 monthly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

32. Primary Outcome: Vital Signs: Heart Rate
Time Frame: from day 1 monthly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

33. Primary Outcome: Vital Signs: Body Temperature
Time Frame: from day 1 monthly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

34. Primary Outcome: Adverse Events
Time Frame: from day 1 weekly to day 365
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

35. Primary Outcome: Genetic Polymorphisms of Fatty Acid Desaturase Genes FADS1 and FADS2
Description: The relation between genetic polymorphisms in the fatty acid desaturase genes Fatty acid desaturase 1 (FADS1) and Fatty acid desaturase 2 (FADS2) and plasma concentrations of linoleic acid, α-linolenic acid, arachidonic acid, docosahexaenoic acid, eicosapentaenoic acid, and Mead acid, as well as relation to and EFAD (triene/tetraene ratio)
Time Frame: once during treatment phase (day 1 to day 365)
Population: as for outcome 1
Arm/Group | Smoflipid | Intralipid, 20%
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected at each study visit until one day after the end of last study treatment (i.e., Study Day 365 in maximum).
Description: There was only one patient treated in the study.
Arm/Group | Smoflipid | Intralipid, 20%
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/0
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Smoflipid (N=1) | Intralipid, 20% (N=0)
BACTERAEMIA (Infections and infestations) | 1 (1) | 0 (0)
HYPOVOLAEMIC SHOCK (Vascular disorders) | 1 (1) | 0 (0)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
FUNCTIONAL GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0)
DEVICE RELATED SEPSIS (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Smoflipid (N=1) | Intralipid, 20% (N=0)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
TACHYCARDIA (Cardiac disorders) | 1 (3) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 1 (1) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0)
LIPASE INCREASED (Investigations) | 1 (1) | 0 (0)
WEIGHT DECREASED (Investigations) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (4) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
METABOLIC ACIDOSIS (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
TETANY (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was released from postmarketing requirement and the product received marketing authorization approval from the U.S. Food & Drug Administration. Therefore, the study was early terminated after treatment of a single patient.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-19): https://cdn.clinicaltrials.gov/large-docs/22/NCT03563222/Prot_SAP_000.pdf